CLINICAL TRIAL: NCT02348866
Title: Bacterial Contamination on Obstetric Resident Surgical Scrubs: a Randomized Trial
Brief Title: Bacterial Contamination on Obstetric Resident Surgical Scrubs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro#00041187
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Bacterial Contamination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): home laundered/home-donned
  Interventions: Other: method of laundering and donning scrubs
- Group 2 (Active Comparator): Hospital laundered/home-donned
  Interventions: Other: method of laundering and donning scrubs
- Group 3 (Active Comparator): Home laundered/hospital donned
  Interventions: Other: method of laundering and donning scrubs
- Group 4 (Active Comparator): Hospital laundered/hospital donned
  Interventions: Other: method of laundering and donning scrubs

INTERVENTIONS:
Other: method of laundering and donning scrubs

SUMMARY:
This study will determine if there is a difference in bacterial contamination (CFU/cm2) between obstetric resident surgical scrubs donned at home and those donned at the hospital.

DETAILED DESCRIPTION:
An area of potential provider-to-patient contamination, and therefore intervention, is in health care worker attire and laundering practices. For providers who work in the operating room or labor & delivery suites, this uniform usually comprises hospital-issued surgical scrubs. To the best of our knowledge, no study has measured the difference in bacterial contamination on surgical scrubs vis-a-vis the two variables most directly affected by hospital policies for surgical attire: site of scrub laundering and site where scrubs were first put on. In addition, no study has measured the prevalence of antibiotic-resistant organisms on surgical scrubs in the obstetric setting. Our primary objective is to measure the difference in bacterial contamination (CFU/cm2) between home-laundered/home-donned scrubs ("home/home," group 1), hospital-laundered/home-donned scrubs ("hospital/home," group 2), home-laundered/hospital-donned scrubs ("home/hospital," group 3), and hospital-laundered/hospital-donned scrubs ("hospital/hospital," group 4) in the obstetric setting. Our secondary objective is to determine the prevalence of antibiotic-resistant organisms on surgical scrubs in the obstetric setting.

ELIGIBILITY:
Inclusion Criteria:

* ob-gyn residents assigned to labor and delivery during the day on one of seven rotation blocks

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
difference in bacterial contamination between scrubs donned at home and those put on in the hospital, when location of laundering is considered (as determined by (CFU/cm2) | 4 days
  4 days of randomization per subject

SECONDARY OUTCOMES:
Prevalence of antibiotic resistant Staphylococcus aureus on surgical scrubs in the obstetric setting | 4 days
  4 days of randomization per subject

CONTACTS AND LOCATIONS:
Overall Officials: Kacey Y Eichelberger, MD, Principal Investigator — Prisma Health-Upstate